CLINICAL TRIAL: NCT04737499
Title: Implementation and Evaluation of A Culturally Tailored Diabetes Self-Management Program for Chinese Americans
Brief Title: Culturally Appropriate Strategies for Chinese Americans With Diabetes (CASCADe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Collaborators: AHMC Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGU IRB#2522
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes
Keywords: Chinese Americans; Type 2 Diabetes; mHealth; Diabetes Self-Management and Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single group pre- and post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CASCADe Intervention (Experimental): Intervention consisted of eight weekly sessions of health education and diabetes management. Topics covered include recognition of diabetes and its complications, risk factors, nutrition knowledge, dietary practices, exercise, behavioral self-monitoring, medication adherence, and stress management. Intervention also included a home visit for training of monitoring devices use, WeChat app and acquiring family support, and weekly WeChat follow-up on education tips, monitoring data summary, and group discussion. The monitoring system used a smartphone to coordinate cloud data transmission from a set of wireless devices to capture daily monitoring data on physical activity, body weight, blood pressure and blood glucose levels.
  Interventions: Behavioral: CASCADe

INTERVENTIONS:
Behavioral: CASCADe — Culturally tailored diabetes self-management and education sessions with mHealth integration

SUMMARY:
The project aimed to evaluate the implementation process and efficacy of a culturally tailored Diabetes Self-Management and Education (DSME) program with mobile health (mHealth) technology integration, entitled Culturally Appropriate Strategies for Chinese Americans with Diabetes (CASCADe), among Chinese American adults with Type 2 diabetes.

DETAILED DESCRIPTION:
The CASCADe program includes 1) a home visit for training of monitoring devices use, WeChat app and acquiring family support, 2) 8 weekly education sessions with a combined format of group class, games, food demonstration, group exercise, video and discussion, 3) WeChat follow-up on education tips, monitoring data summary, and group discussion. The monitoring system used a smartphone to coordinate cloud data transmission from a set of wireless devices to capture daily monitoring data on physical activity, body weight, blood pressure and blood glucose levels. WeChat app was used to facilitate behavioral self-monitoring by providing daily messages related to diabetes education curriculum, weekly summary reports on monitoring data as well as reinforcement messages and group discussion on readings and monitoring results implication. A single group pre-post-test design was adopted to evaluate changes of primary (HbA1c) and secondary (Self-efficacy, quality of life and stress coping) outcomes assessed at pre and post of intervention. Engagement and adherence in education sessions and self-monitoring system, and satisfaction with the content and delivery of intervention were also evaluated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* have been diagnosed with Type 2 diabetes
* having been managing diabetes with diet, oral hypoglycemic agents or insulin, or both
* confirmed HbA1c level >=6.5% and <10%
* 21-75 years old
* residents of San Gabriel Valley
* speak and understand of Mandarin
* willing to use the smartphone-based monitoring devices provided by the project.

Exclusion Criteria:

* unable or unwilling to give informed consent
* plan to move out of the area within the 1-year participation study period
* are or plan to be pregnant or breastfeeding in the next 12 months
* have a condition that inhibits movement (e.g., unable to walk unaided, or cannot walk 1/4 mile without stopping)
* have major physical disability or condition that prevents them from participating in person.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Change of Concentration of HbA1c | Change from baseline HbA1c at 3 months
  HbA1c was assessed using the testing kit of A1C Now+ with a finger prick of blood by trained data collector.

SECONDARY OUTCOMES:
Change of Score of Self-efficacy | Change from baseline Self-efficacy score at 3 months
  Chinese version of diabetes self-management self-efficacy scale included 20 items with likert-like response scale of 1-5 and minimum score of 20 and maximum score of 100.
Change of Score of Quality of life | Change from baseline Quality of life score at 3 months
  Chinese version of diabetes quality of life scale included 15 items with likert-like response scale of 1-5, and minimum score of 15 and maximum score of 75. .

CONTACTS AND LOCATIONS:
Locations (1):
- Clarement Graduate University, Claremont, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets with individual participant data will be provided by the Principal Investigator upon request. All data sharing requests will be reviewed and approved by the Office of Research and Sponsored Programs at Claremont Graduate University and the research investigating team.

REFERENCES:
- [Derived] Xie B, Li Y, Hwang WC, Niu Z, Lei X, Yu R, Lai Y, Fong T, Ma Y. A Culturally Tailored Diabetes Self-Management Education Program With Mobile Health Integration for Chinese Americans With Type 2 Diabetes: Development and Pilot Evaluation Study. JMIR Form Res. 2026 Feb 3;10:e77372. doi: 10.2196/77372. PMID 41632517